CLINICAL TRIAL: NCT01347463
Title: Validation of the Ipsilateral Nipple as the Directional Guide for Internal Jugular Vein (IJV) Catheterization
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Assistant professor, Seoul National University Hospital
Other Study IDs: IJV-cath-nipple
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Ipsilateral Nipple; Internal Jugular Vein; Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Traditional
  Interventions: Procedure: SCM triangle - ipsilateral nipple

INTERVENTIONS:
Procedure: SCM triangle - ipsilateral nipple — draws the tract of the IJV using the SCM triangle head and the ipsilateral nipple

SUMMARY:
Traditional teaching that suggests the ipsilateral nipple as the directional guide for needle advancement during Internal Jugular Vein (IJV) catheterization has weak grounds.

The investigators attempt to validate this long-standing statement.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over the age of 18 undergoing general anesthesia

Exclusion Criteria:

* history of neck or breast surgery
* anatomical anomaly of the neck or breast
* neck mass
* breast mass

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled to undergo general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
difference in angle | 1 day
  difference in angle between traditional (triangular head of the SCM - ipsilateral nipple) and ultrasound guided tract

CONTACTS AND LOCATIONS:
Locations (1):
- Boramae Medical Center, Seoul, South Korea